CLINICAL TRIAL: NCT01547416
Title: The Effect of Combined General/Epidural Anesthesia Versus General Anesthesia on Diaphragmatic Function After Robot-assisted Prostatectomy
Brief Title: The Effect of Combined General/Epidural Anesthesia Versus General Anesthesia on Diaphragmatic Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0344
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: Diaphragmatic dysfunction; General anesthesia; Epidural Anesthesia
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections, Epidural; Ropivacaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- combined general/epidural anesthesia (Experimental): epidural catheter was inserted in group GE at T8/9, T9/10, or T10/11 interspinous space with a 17-gauge Tuohy needle in lateral decubitus position and advanced 5 cm cephalad. Epidural analgesia was maintained using the patient-controlled analgesia technique.
  Interventions: Drug: epidural 250mL of 0.2% ropivacaine and 2 μg/mL of fentanyl, 5 mL/hr continuous infusion and 0.5 mL bolus dose
- General anesthesia (Active Comparator): Patients allocated to general anesthesia group did not receive epidural anesthesia.
  Interventions: Drug: no epidural drug administered

INTERVENTIONS:
Drug: epidural 250mL of 0.2% ropivacaine and 2 μg/mL of fentanyl, 5 mL/hr continuous infusion and 0.5 mL bolus dose — Before the induction of anesthesia, epidural catheter was inserted in group GE at T8/9, T9/10, or T10/11 interspinous space with a 17-gauge Tuohy needle in lateral decubitus position and advanced 5 cm cephalad. .
  Epidural analgesia was maintained using the patient-controlled analgesia technique containing 250 mL of 0.2% ropivacaine and 2 μg/mL fentanyl with setting of 5 mL/hr for continuous infusion and 0.5 mL of bolus dose. Lockout time was set to 15 min.
  General anesthesia was induced with 2 mg/kg of propofol and 50 mg of rocuronium. After tracheal intubation, anesthesia was maintained with sevoflurane. All the patients were ventilated with controlled mode of 8 mL/kg of ideal body weight and respiratory rate was adjusted to maintain end-tidal carbon dioxide between 35-40 mmHg.
  Arms: combined general/epidural anesthesia
Drug: no epidural drug administered — Patients allocated to general anesthesia group and DID NOT receive epidural anesthesia.
  General anesthesia was induced with 2 mg/kg of propofol and 50 mg of rocuronium. After tracheal intubation, anesthesia was maintained with sevoflurane. All the patients were ventilated with controlled mode of 8 mL/kg of ideal body weight and respiratory rate was adjusted to maintain end-tidal carbon dioxide between 35-40 mmHg.
  Arms: General anesthesia

SUMMARY:
The aim of this study was to investigate whether robot assisted laparoscopic radical prostatectomy give rise to the impairment of diaphragmatic function postoperatively, and whether combined general/epidural anesthesia could provide better postoperative diaphragmatic function.

DETAILED DESCRIPTION:
Diaphragmatic dysfunction after abdominal surgery can result in extended hospital stay and increased medical costs, because it is related with atelectasis, lung collapse or pneumonia. The mechanism of diaphragm dysfunction is thought to be from not only direct injury to abdominal wall and viscera but inhibitory reflexes of phrenic activity. Thoracic or upper abdominal surgery is suggested as a risk factor of postoperative diaphragm dysfunction, and perioperative analgesic modality is also known to affect diaphragm movements. But there has been no trial to investigate the effect of laparoscopic pelvic surgery such as prostatectomy on diaphragm movement. Moreover, it is not clear if minimally invasive Robot-assisted laparoscopic radical prostatectomy (RALRP) has any influence on respiratory and diaphragm functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients of over 18 years of age undergoing elective Robot-assisted laparoscopic radical prostatectomy

Exclusion Criteria:

* Patients with previous history of smoking, cardiopulmonary or neuromuscular disease or obesity (body mass index > 30 kg.m-2)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of diaphragm movement using sonography (diaphragm inspiratory amplitude, diaphragm inspiratory and expiratory velocity)on postoperative day 1 and 2 from baseline (day before surgery) | on the day before surgery until postoperative day 2
  The measurements of diaphragmatic motion were attained at the posterior surface of the diaphragm. From the tracings on M-mode, the distance between echogenic lines (DIA) in cm and diaphragm inspiratory/expiratory velocity in cm.s-1 during quiet, deep, and sniff breathing were measured on the frozen images. Three consecutive sonographic examinations were performed, and the highest value of three measurements was recorded

SECONDARY OUTCOMES:
Change in pulmonary function test on postoperative day 1 and 2 from baseline (day before surgery) | on the day before surgery until postoperative day 2
  Spirometric measurements included vital capacity (VCIN), forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC, peak expiratory flow rate (PEF), maximal midexpiratory flow rate (MMEF), tidal volume (VT), and expiratory residual volume (ERV)

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, M.D. Ph.D., Principal Investigator — Severance Hospital, Yonsi University Health System
Locations (1):
- Severence Hospital, Yonsei University Health System, Seoul, South Korea